CLINICAL TRIAL: NCT01878994
Title: Evaluation of Family Intervention Program for the Treatment of Overweight or Obese Children (Nereu Program): Randomized Clinical Trial
Brief Title: Evaluation of a Family Intervention Program for the Management of Overweight or Obese Children
Acronym: NEREU
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Associació NEREU (Unknown); INEFC-Lleida (Other); USR-ICS. Atenció Primària Lleida (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PI12/02220
Record Dates: First submitted 2013-06-11; First posted 2013-06-17 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2013-06

CONDITIONS: Overweight; Obesity; Children
Keywords: Overweight; Obesity; Children; Behaviour; Physical Activity; Nutrition
MeSH Terms: conditions — Overweight; Obesity; Behavior; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Counselling Group (Placebo Comparator): Each family will receive a single monthly meeting, a total of 8 with 10 minutes duration each one. The sessions will take place in the consultation of the paediatrician and it will be delivered by the child's nurse or/and paediatrician. The sessions' contents are about promotion of healthy eating and physical activity habits.
  Interventions: Behavioral: Counselling group
- Nereu Group (Experimental): The Nereu treatment program is an intensive family-based behavioural multi-component lifestyle intervention. Consist in an intensive treatment of 8 months duration (from October to May, that is, an academic year). The intervention is a multidisciplinary intervention consisting in 4 structured components: (a) physical activity training for children, (b) family theoretical and practical sessions for parents, (c) behaviour strategies, that involves both parental and child participation (d) weekend extra activities.
  Interventions: Behavioral: Nereu group

INTERVENTIONS:
Behavioral: Counselling group
  Arms: Counselling Group
Behavioral: Nereu group
  Arms: Nereu Group

SUMMARY:
Objectives: To evaluate the effectiveness of the Nereu program compared to standard care (advice on increased physical activity and nutrition) such as a health intervention tool for the childhood obesity management

Methods/Design: The study design is a randomized controlled multicenter clinical trial using two types of treatment. Population and sample: Children 6 to 12 years with overweight or obesity, according to the z score of body mass index (BMI z) >= 1 for age and gender defined by International Obesity Task Force (IOTF). It is considered necessary to recruit 100 children: 50 control group (CG) and 50 Intervention (IG). Study Intervention: Nereu Group: 8 month intervention with 3 weekly training sessions doing physical exercise for children and a weekly session for parents of physical activity and healthy eating habits and behaviour strategies, that involves both parental and child participation. The control group will receive a monthly session of healthy physical and eating habits. Main Outcome Measures: Improvement of BMI z, physical activity and nutrition habits, behaviour components and quality life related to health at the end, 6 and 12 months after intervention.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 6 to 12 years old
* Overweight or obese according to the IOTF criteria

Exclusion Criteria:

* Medical co-morbidities: Diabetes mellitus or hypercholesterolemia or cardiovascular disease that could be contraindicate the sport practice.
* Use of medication that might have an effect on weight loss.
* previous enrolment in another similar treatment program based on reducing obesity.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-06 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Body mass index z score (BMIz) | 4 times: at baseline, at the end of the intervention (8 months later of the baseline), 6 and 12 months post intervention
  Weight is measured to the nearest of 0.1 kg using an electronic scale and height (Ht) to the nearest of 0.1 cm with a stadiometer, in lightly dressed and without shoes. The BMIz is calculated according z score of BMI adjusted by age and gender (IOTF).

SECONDARY OUTCOMES:
Change from baseline in Physical activity habits | 4 times: at baseline, at the end of the intervention (8 months later of the baseline), 6 and 12 months post intervention
  To measure physical activity will be used an Actigraph accelerometers (GT3X+ models), it will be wear by participants during all day for seven consecutive days.

CONTACTS AND LOCATIONS:
Overall Officials: Noemí Serra, Principal Investigator — INEFC-LLEIDA, University of Lleida; Concepció Teixidó, Principal Investigator — Institut Català de la Salut - Atenció primaria - Lleida
Locations (1):
- USR- Lleida. Atenció primaria. IDIAP Jordi Gol, Lleida, Lleida, Spain

REFERENCES:
- [Derived] Serra-Paya N, Ensenyat A, Castro-Vinuales I, Real J, Sinfreu-Bergues X, Zapata A, Mur JM, Galindo-Ortego G, Sole-Mir E, Teixido C. Effectiveness of a Multi-Component Intervention for Overweight and Obese Children (Nereu Program): A Randomized Controlled Trial. PLoS One. 2015 Dec 14;10(12):e0144502. doi: 10.1371/journal.pone.0144502. eCollection 2015. PMID 26658988
- [Derived] Serra-Paya N, Ensenyat A, Real J, Castro-Vinuales I, Zapata A, Galindo G, Sole-Mir E, Bosch-Munoz J, Mur JM, Teixido C. Evaluation of a family intervention programme for the treatment of overweight and obese children (Nereu Programme): a randomized clinical trial study protocol. BMC Public Health. 2013 Oct 23;13:1000. doi: 10.1186/1471-2458-13-1000. PMID 24153001